CLINICAL TRIAL: NCT07058987
Title: A Prospective Randomized Controlled Study on the Effects of Enhanced External Counterpulsation Combined With Cardiac Rehabilitation on Cardiac Function and Exercise Capacity in Patients With Atrial Fibrillation
Brief Title: Effects of Enhanced External Counterpulsation Combined With Cardiac Rehabilitation in Patients With Atrial Fibrillation
Acronym: EECP AF CR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Xiaowei Zhang, lanzhou university second hospital, Lanzhou University Second Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LZUSH-AFCR-2025-001; lanzhou university (Other: lanzhou university second hospital)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF); Heart Failure (HF); Cardiac Rehabilitation
Keywords: Atrial Fibrillation; Cardiac Rehabilitation; Enhanced External Counterpulsation; Exercise Capacity
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Cardiac Rehabilitation; Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group (receiving EECP combined with cardiac rehabilitation) or the control group (receiving routine medical care). Each participant will remain in their assigned group throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EECP + Cardiac Rehabilitation (Experimental): Participants will receive enhanced external counterpulsation (EECP) plus a structured cardiac rehabilitation program that includes individualized aerobic exercise training, health education, psychological support and lifestyle counselling.
  Interventions: Behavioral: Cardiac Rehabilitation Combined With EECP
- Routine Medical Care (Active Comparator): Participants will continue to receive standard pharmacologic management and routine clinical follow-up for atrial fibrillation without EECP or formal cardiac rehabilitation.
  Interventions: Other: Routine Medical Care

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation Combined With EECP — This intervention consists of a comprehensive cardiac rehabilitation program that includes individualized aerobic exercise training, health education, psychological support, and lifestyle counseling, combined with enhanced external counterpulsation (EECP) therapy administered according to standard cardiovascular protocols. The combined intervention is designed to improve cardiac function, exercise tolerance, and quality of life in patients with atrial fibrillation.
  Other Names: Enhanced External Counterpulsation; EECP; Cardiac Rehabilitation; CR; Lifestyle Modification; Exercise Training
  Arms: EECP + Cardiac Rehabilitation
Other: Routine Medical Care — Participants in the control group will receive standard medical treatment for atrial fibrillation as prescribed by their attending physicians, without enhanced external counterpulsation or structured cardiac rehabilitation. This may include pharmacological therapy, routine clinical monitoring, and general lifestyle advice.
  Other Names: Standard Care; Usual Care; Pharmacological Management
  Arms: Routine Medical Care

SUMMARY:
This is a prospective randomized controlled trial designed to evaluate the effectiveness of enhanced external counterpulsation (EECP) combined with cardiac rehabilitation in patients with atrial fibrillation. The study aims to assess whether this combined intervention can improve cardiac function and exercise capacity compared to standard care alone. Eligible participants will be randomly assigned to receive either the EECP plus cardiac rehabilitation program or routine treatment. Primary outcomes include changes in left ventricular ejection fraction (LVEF) and six-minute walking distance (6MWD). The study will be conducted at Lanzhou University Second Hospital.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common cardiac arrhythmia associated with impaired ventricular function, reduced exercise tolerance, and increased risk of cardiovascular events. While pharmacological treatments and catheter ablation are widely used, non-pharmacological interventions such as enhanced external counterpulsation (EECP) and cardiac rehabilitation (CR) may offer additional benefits for improving cardiac performance and quality of life. This prospective, single-center, randomized controlled trial aims to evaluate the effects of EECP combined with a structured cardiac rehabilitation program in patients with persistent or paroxysmal atrial fibrillation. A total of approximately 200 eligible participants will be randomized in a 1:1 ratio to receive either EECP plus cardiac rehabilitation (intervention group) or routine medical care (control group) for a defined treatment period. The cardiac rehabilitation program will include individualized exercise training, health education, risk factor management, and follow-up support. EECP will be performed according to standard protocols for cardiovascular patients. Primary outcome measures will include changes in left ventricular ejection fraction (LVEF) and six-minute walking distance (6MWD) from baseline to the end of the intervention. Secondary outcomes may include assessments of quality of life, symptoms, and biomarkers. Safety and feasibility will also be recorded. This study is expected to provide clinical evidence supporting the integration of EECP and cardiac rehabilitation as a non-invasive, multidimensional treatment approach in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years
* Diagnosed with persistent or paroxysmal atrial fibrillation, confirmed by ECG or Holter
* Stable medical condition and able to participate in cardiac rehabilitation and EECP therapy
* Provided written informed consent

Exclusion Criteria:

* Recent acute myocardial infarction, unstable angina, or decompensated heart failure within the past 4 weeks
* Severe valvular heart disease or left ventricular ejection fraction <30%
* Severe peripheral vascular disease or deep vein thrombosis
* Severe pulmonary disease or active infection
* History of bleeding disorders or contraindications to EECP
* Cognitive impairment or psychiatric condition affecting study participation
* Participation in another clinical trial within the past 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) from Baseline to Week 12 | Baseline and 12 weeks after intervention
  LVEF will be assessed using transthoracic echocardiography to evaluate improvement in systolic cardiac function.

SECONDARY OUTCOMES:
Change in 6-Minute Walk Distance (6MWD) | Baseline and 12 weeks
  6MWD will be measured to assess changes in functional exercise capacity.
Incidence of Adverse Events | Throughout the 12-week intervention period
  All adverse events related to EECP or cardiac rehabilitation will be recorded to assess safety and tolerability.
Change in NT-proBNP Level | Baseline and 12 weeks
  Blood samples will be collected to assess changes in NT-proBNP, a biomarker of cardiac stress and heart failure severity.
Change in Health-Related Quality of Life (HRQoL) Measured by SF-36 Total Score | Baseline and 12 weeks
  The validated Chinese version of the Short-Form 36 Health Survey (SF-36; total score range 0 - 100, with higher scores indicating better health status) will be administered face-to-face by trained study nurses at baseline and Week 12. The primary metric will be the change in total SF-36 score computed using the standard scoring algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei Zhang PhD, Principal Investigator — Lanzhou University Second Hospital
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided